CLINICAL TRIAL: NCT00965770
Title: Preventing Repeat Abortion: Is the Immediate Insertion of Intrauterine Devices Post-abortion a Cost-effective Option Associated With Fewer Repeat Abortions? Findings From 2001-2004 Data
Brief Title: Post Abortion IUD & Recurrent Abortion 2001-2004
Status: Terminated | Type: Observational
Why Stopped: This study is a retrospective chart review study, not a clinical trial.
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Wendy Norman, Principle Investigator, University of British Columbia
Other Study IDs: H09-01871
Record Dates: First submitted 2009-08-24; First posted 2009-08-26 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Abortion Rate
Keywords: abortion; intrauterine device; cost-effectiveness
MeSH Terms: interventions — Intrauterine Devices

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- IUD: Repeat abortion rate in women receiving IUDs immediately post-abortion
  Interventions: Device: Intrauterine device (IUD)

INTERVENTIONS:
Device: Intrauterine device (IUD) — Women choosing to have an intrauterine device (IUD) inserted immediately post-abortion

SUMMARY:
It has been shown that the immediate insertion of intrauterine devices (IUDs) post-abortion prevents repeat abortions. The researchers hypothesize that providing free IUDs post-abortion will be associated with a lower rate of repeat abortion in a Canadian population. Further, the researchers hypothesize that providing free IUDs post-abortion will be associated with decreased costs for the health care system.

DETAILED DESCRIPTION:
The researchers intend to demonstrate whether there are statistically significant differences in the rates of repeat abortions between three groups: 1. women choosing to have an intrauterine device (IUD) inserted immediately post-abortion, 2. those choosing to begin oral contraceptives immediately post-abortion, and 3. all other choices for post abortion contraception including those stating an intention to obtain contraceptives at a later time or from an alternate location or to use no contraception. This data will then be used to conduct a cost-effectiveness analysis of health system provision for cost-free IUDs post-abortion.

The researchers will conduct a retrospective observational cohort study by chart review. The researchers propose to review the charts of 600 women undergoing abortions between January 1, 2001 and December 31, 2004 at Kelowna General Hospital's Women's Services Clinic. The researchers will record the following data from each chart: age, parity, gestational age, date of index therapeutic abortion (TA), dates of subsequent TAs, contraception used at the time of the index conception, contraceptive method chosen post-abortion, and outcome of follow-up at two weeks, such as expulsion of IUD. The researchers will also record the recurrent pregnancy rates.

ELIGIBILITY:
Inclusion Criteria:

* Female resident of Interior Health region seeking an abortion between January 1, 2001 and December 31, 2004

Exclusion Criteria:

* Women undergoing abortions for fetal genetic abnormalities

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female resident of Interior Health region seeking an abortion
Sampling Method: Non-Probability Sample
Enrollment: 1101 (Actual)
Dates: Start 2011-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
The proportion of repeat abortions at five years from the index abortions. | 5 years

SECONDARY OUTCOMES:
A cost-effectiveness analysis of providing free IUDs to women immediately post-abortion; correlation of repeat and index abortions with obstetrical, demographic and contraceptive history factors. | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Norman, Dr., Principal Investigator — University of British Columbia
Locations (1):
- Women's Services Clinic, Kelowna General Hospital, Kelowna, British Columbia, Canada